CLINICAL TRIAL: NCT06804421
Title: Late Neurological Ischemic Deficit in Patients Suffering From Subarachnoid Hemorrhage: Diagnosis and Treatment
Brief Title: Diagnosis and Treatment of Late Neurological Ischemic Deficit in Patients Suffering From Subarachnoid Hemorrhage.
Acronym: DINTESA
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS San Gerardo dei Tintori (Other)
Responsible Party: Sponsor
Other Study IDs: DINTESA (4533)
Record Dates: First submitted 2025-01-20; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Aneurysmal Subarachnoid Haemorrhage; Delayed Ischemic Neurological Deficit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- aSAH group: Patients diagnosed with aneurysmal subarachnoid hemorrhage.
- DIND group: Patients diagnosed with aneurysmal subarachnoid hemorrhage who develop delayed ischemic neurologic deficit.

SUMMARY:
Recent studies state that patients affected by aneurysmal subarachnoid hemorrhage (aSAH) today survive longer because they are treated early. Unfortunately, patients often develop chronic disabling neurological deficits at a rate that is still unacceptable given the progress in the specific treatment of this pathology and the volume of systems of neurological monitoring available to date in Italy.

The main cause of unfavorable neurological outcome is delayed cerebral ischemia (DCI), often resulting from symptomatic vasospasm defined as delayed neurological ischemic deficit (DIND). The incidence of DIND is not defined and is difficult to diagnose early as there is no gold standard for identifying it, nor guidelines regarding the most effective treatment.

Given these gaps, the primary objective of this study is to describe the incidence of DIND in patients affected by aSAH, collecting information regarding the diagnostic imaging (neurological symptom on clinical examination or alteration on instrumental monitoring). Secondary objectives will be to evaluate the different therapeutic strategies adopted in the different participating centers and compare these strategies to mortality and short- and long-term functional neurological outcome. Furthermore, as there are no data in the literature, the Investigators want to describe the indications, usefulness and intensity of treatment in the aSAH patient in case of monitoring of parenchymal intracranial pressure.

DETAILED DESCRIPTION:
Aneurysmal subarachnoid hemorrhage (aSAH) is a particular form of hemorrhagic stroke characterized by blood spillage into the intracranial subarachnoid spaces due to the rupture of an aneurysm of a large cerebral arterial vessel of the circle of Willis. It can cause sudden and intense symptoms, such as violent headache, nausea, vomiting, neck stiffness and sensitivity to light, but also loss of consciousness, cardiac arrest and death.

The pre-hospital mortality rate in the literature remains high (22-26%), even if it is lower than in previous decades. However, the number of patients discharged from hospital with permanent disabilities is increasing, especially those of working age (the average age at onset of symptoms is 55 years), contributing significantly to public health costs.

The incidence of aSAH worldwide is approximately 6.1 cases per 100,000 people per year, but there are national differences. In Italy, for example, it is 11.2 (10.5-12.4) cases per 100,000 inhabitants per year.

At the onset of symptoms, once the aneurysmal origin of the cerebral hemorrhage has been confirmed through radiological examinations, it is essential to promptly ensure treatment of the ruptured aneurysm. Early repair of the ruptured aneurysm is recommended within 24 to 72 hours, via endovascular coiling or neurosurgical clipping. This allows to prevent any rebleeding and reduce the risk of cerebral vasospasm, as it reduces the amount of blood distributed in the subarachnoid space. The latter, in fact, represents the main inflammatory stimulus on large cerebral arteries, favoring the vasoconstriction reaction which manifests itself angiographically and/or ultrasonographically in 70% of cases. Cerebral vasospasm is very often clinically silent, since the reduction of the vascular lumen is not sufficient to generate the conditions of discrepancy between the arterial flow of the perfused brain parenchyma and its metabolic demand.

However, in 20-30% of cases a neurological deterioration also occurs, called delayed ischemic neurological deficit or DIND (Delayed Ischemic Neurological Deficit), defined as a focal neurological deterioration (appearance of at least one of the symptoms including hemiparesis, aphasia, hemianopsia or neglect) or global (sudden neurological worsening leading to at least a two-point decrease in the Glasgow Scale or the appearance of anisocoria or pupillary reactivity). DIND is not always immediately evident after securing the aneurysm, and it is necessary to exclude other causes of neurological deterioration, such as hydrocephalus, convulsions, rebleeding and hyponatremia in order to confirm it.

Identifying DIND early is essential to prevent the formation of a true ischemic core in the area affected by vasospasm, i.e. late cerebral ischemia, DCI (Delayed Cerebral Ischemia), defined by radiological criteria: evidence of cerebral infarction on brain computed tomography (CT) scan or brain magnetic resonance imaging (MRI) within 6 weeks of onset of aSAH complicated by vasospasm.

DIND, in fact, is the main preventable cause of unfavorable neurological-functional outcome and DCI in patients with SAH.

Regarding the identification of DIND, it is certainly crucial to carry out a systematic clinical neurological examination on the awake patient. In comatose patients, or in those in whom it is not possible to carry out a sedation window, multimodal instrumental monitoring is certainly helpful. In fact, if the patient is sedated or cannot be awakened, the information deriving from the inspection (pupillary reactivity and isocoria) should be integrated with continuous electroencephalographic monitoring (cEEG) and/or transcranial color Doppler ultrasound (TCD)ccc. Instrumental monitoring is, in fact, fundamental in those patients in whom a suspension of sedation generates an increase in intracranial pressure and consequent reduction in cerebral oxygenation, making clinical neurological evaluation impossible.

The alterations associated with DIND most commonly described during quantitative EEG (qEEG) are decreased alpha/delta ratio and reduced alpha variability. EEG changes may precede clinical deterioration by several hours, and allow for a differential diagnosis with nonconvulsive status epilepticus. Instrumental vasospasm is defined as an average blood flow velocity > 120 cm/sec detected ultrasonographically via TCD. Instead, clinical vasospasm, i.e. DIND that requires treatment, is diagnosed in case of speed of at least 200 cm/sec, or increased by 50 cm/sec in the last 24 hours, or even if the Lindeegard index is greater of 3 (defined as the ratio of flow velocities between the middle cerebral artery and the ipsilateral distal internal carotid artery, MCA/ICA).

Regarding second-level tests, in sedated or unconscious patients, it is also reasonable to perform screening through repeated imaging tests, such as computed perfusion tomography (CTP), cerebral angiotomography (CTA) and intracranial vessel angiography ( TSA). The use of CTP is increasingly widespread: it detects imminent ischemia by decreasing cerebral perfusion, thus identifying salvageable brain tissue (ischemic penumbra) before irreversible brain damage occurs. This approach, however, involves transporting the critically ill patient to radiology and administering a contrast medium, adding considerable risks. It should also be underlined that, in case of clinical or instrumental suspicion of DIND, in some centers second level tests are used less and less, intervening early with therapy to resolve it.

As with the diagnostic procedure, the therapeutic strategies implemented are also very different from each other, and none has been proven to be more effective than another. They can be more or less invasive, and the main ones are:

* hemodynamic therapy, i.e. permissive hypertension, in which systemic blood pressure is increased to increase cerebral perfusion and ensure that an adequate quantity of blood supplies the brain parenchyma downstream of vasospasm;
* local intra-arterial pharmacological therapy, in bolus or continuous infusion, with a vasodilator drug (calcium antagonist/milrinone);
* mechanical therapy, whereby action is taken on the muscular wall of the vessel in question by carrying out angioplasty with a transluminal balloon.

Innovative techniques, such as stent retriever angioplasty, which also allows the application of intra-arterial calcium channel antagonists, can be an additional tool in selected patients with refractory vasospasm.

To date, there is no gold standard for diagnosing DIND, evidence on which patients are at greatest risk of developing it and recommendations regarding the most effective treatment to resolve it. Management is delegated to the multidisciplinary department team of each centre.

In conclusion, also in light of the recent guidelines on aSAH, it is urgent to establish how to prevent DCI, identifying the onset of DIND early, both clinically and instrumentally.

With this study the Investoigators aim to determine the incidence of DIND in patients with aSAH, to evaluate the effectiveness of different treatments and to compare the different diagnostic/therapeutic strategies in the participating centers, investigating the impact of DIND on short-term and long-term neurological-functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Primary diagnosis of subarachnoid hemorrhage due to rupture of a cerebral artery aneurysm confirmed by cerebral angiotomography or angiography of the intracranial vessels, with the need for admission to the Intensive Care Unit
* Signing the Informed Consent form to participate in the study according to current local regulations.

Exclusion Criteria:

* Age < 18 years
* Primary diagnosis of subarachnoid hemorrhage sine materia, i.e. post-traumatic or caused by arteriovenous malformation or bleeding from a brain tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The enrolling centers are mainly located in the Lombardy region, Italy. All Lombard and selected national (from other regions) centers with neurosurgery were involved.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2024-09-28 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
DIND incidence | 12 months
  Describe the incidence of DIND in patients affected by aSAH. The presence of a suspicious alteration for DIND at the neurological clinical examination (if the patient is awake or if a sedation window is possible) or instrumental (if the clinical examination is not possible), confirmed or not by radiological examinations, will be recorded.

SECONDARY OUTCOMES:
Imaging application | 12 months
  Describe and analyze the variability of the diagnostic methods (clinical and instrumental examination) applied by each center to identify DIND in patients with aSAH and how this is treated.
Neurological-functional outcome assessment | 12 months
  Evaluate the impact of DIND and its treatment on short-term and long-term neurological-functional outcomes by mortality at 6 months and 12 months after the acute event.
Invasive monitoring of intracranial pressure | 12 months
  To evaluate the usefulness of invasive monitoring of intracranial pressure (ICP) in guiding the treatment of patients with SAH by comparing the variation of intracranial pressure in patients who have ICP monitoring with the intensity of the treatment applied (TIL, Therapy Intensity Level).
Neurological-functional outcome assessment | 12 months
  Evaluate the impact of DIND and its treatment on short-term and long-term neurological-functional outcomes by neurological-functional outcome (GOSE, Glasgow Outcome Scale Extended) at 6 months and 12 months after the acute event. From GOSE=1 (death) to GOSE=8 (good recovery).
Neurological-functional outcome assessment | 12 months
  Evaluate the impact of DIND and its treatment on short-term and long-term neurological-functional outcomes by neurological-functional outcome (mRS, modified Rankin Scale) at 6 months and 12 months after the acute event. From mRS=0 (no symptoms) to mRS=5 (severe disability).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Citerio, Professor, Head od Department, Principal Investigator — Fondazione IRCCS San Gerardo dei Tintori - Monza, Italy
Locations (33):
- Italy (33):
  - ASST Papa Giovanni XXIII, Bergamo, BG
  - IRCCS Istituto delle Scienze Neurologiche, Bologna, BO
  - ASST Spedali Civili, Brescia, BS
  - Fondazione Poliambulanza, Brescia, BS
  - ASST Lariana Ospedale Sant'Anna, San Fermo della Battaglia, CO
  - ASST Cremona, Cremona, CR
  - Azienda Ospedaliero-Universitaria Careggi, Florence, FI
  - IRCCS Ospedale Policlinico San Martino, Genova, GE
  - ASST Lecco - Ospedale A. Manzoni, Lecco, LC
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, MB
  - ASST Ovest Milanese - Ospedale di Legnano, Legnano, MI
  - ASST Fatebenefratelli Sacco, Milan, MI
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, MI
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - ASST Santi Paolo e Carlo - Ospedale San Carlo Borromeo, Milan, MI
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, MI
  - Human Research Hospital, Rozzano, MI
  - IRCCS San Raffaele, Segrate, MI
  - ASST Mantova, Mantova, MN
  - Azienda Ospedale-Università di Padova, Padua, PD
  - Azienda Ospedaliera di Perugia, Perugia, PG
  - Azienda Ospedaliero-Universitaria di Parma, Parma, PR
  - Fondazione IRCCS Policlinico San Matteo, Pavia, PV
  - Azienda Ospedaliera San Camillo Forlanini, Roma, RM
  - Fondazione Policlinico Universitario A. Gemelli, Roma, RM
  - ASST Valtellina e Alto Lario, Sondrio, SO
  - ASL Città di Torino - Ospedale San Giovanni Bosco, Torino, TO
  - Azienda Sanitaria Universitaria Giuliano Isontina, Trieste, TS
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine, UD
  - ASST Sette Laghi - Ospedale di Circolo e Fondazione Macchi, Varese, VA
  - Ospedale San Bortolo, Vicenza, VI
  - Azienda Ospedaliero Universitaria Integrata, Verona, VR
  - AOU Maggiore della Carità, Novara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Su YS, Ali MS, Pukenas BA, Favilla CG, Zanaty M, Hasan DM, Kung DK. Novel Treatment of Cerebral Vasospasm Using Solitaire Stent Retriever-Assisted Angioplasty: Case Series. World Neurosurg. 2020 Mar;135:e657-e663. doi: 10.1016/j.wneu.2019.12.097. Epub 2019 Dec 24. PMID 31881345
- [Result] Rass V, Helbok R. How to diagnose delayed cerebral ischaemia and symptomatic vasospasm and prevent cerebral infarction in patients with subarachnoid haemorrhage. Curr Opin Crit Care. 2021 Apr 1;27(2):103-114. doi: 10.1097/MCC.0000000000000798. PMID 33405414
- [Result] Yamaki VN, Cavalcanti DD, Figueiredo EG. Delayed Ischemic Neurologic Deficit after Aneurysmal Subarachnoid Hemorrhage. Asian J Neurosurg. 2019 Jul-Sep;14(3):641-647. doi: 10.4103/ajns.AJNS_15_19. PMID 31497080
- [Result] Vergouwen MD, Vermeulen M, van Gijn J, Rinkel GJ, Wijdicks EF, Muizelaar JP, Mendelow AD, Juvela S, Yonas H, Terbrugge KG, Macdonald RL, Diringer MN, Broderick JP, Dreier JP, Roos YB. Definition of delayed cerebral ischemia after aneurysmal subarachnoid hemorrhage as an outcome event in clinical trials and observational studies: proposal of a multidisciplinary research group. Stroke. 2010 Oct;41(10):2391-5. doi: 10.1161/STROKEAHA.110.589275. Epub 2010 Aug 26. PMID 20798370
- [Result] Wilson CD, Shankar JJ. Diagnosing Vasospasm After Subarachnoid Hemorrhage: CTA and CTP. Can J Neurol Sci. 2014 May;41(3):314-9. doi: 10.1017/s031716710001725x. PMID 24718816
- [Result] Wahood W, Rizvi AA, Alexander AY, Yolcu YU, Lanzino G, Brinjikji W, Rabinstein AA. Trends in Admissions and Outcomes for Treatment of Aneurysmal Subarachnoid Hemorrhage in the United States. Neurocrit Care. 2022 Aug;37(1):209-218. doi: 10.1007/s12028-022-01476-5. Epub 2022 Mar 18. PMID 35304707
- [Result] Krishnamurthi RV, Ikeda T, Feigin VL. Global, Regional and Country-Specific Burden of Ischaemic Stroke, Intracerebral Haemorrhage and Subarachnoid Haemorrhage: A Systematic Analysis of the Global Burden of Disease Study 2017. Neuroepidemiology. 2020;54(2):171-179. doi: 10.1159/000506396. Epub 2020 Feb 20. PMID 32079017
- [Result] Claassen J, Park S. Spontaneous subarachnoid haemorrhage. Lancet. 2022 Sep 10;400(10355):846-862. doi: 10.1016/S0140-6736(22)00938-2. Epub 2022 Aug 16. PMID 35985353
- [Result] Hoh BL, Ko NU, Amin-Hanjani S, Chou SH-Y, Cruz-Flores S, Dangayach NS, Derdeyn CP, Du R, Hanggi D, Hetts SW, Ifejika NL, Johnson R, Keigher KM, Leslie-Mazwi TM, Lucke-Wold B, Rabinstein AA, Robicsek SA, Stapleton CJ, Suarez JI, Tjoumakaris SI, Welch BG. 2023 Guideline for the Management of Patients With Aneurysmal Subarachnoid Hemorrhage: A Guideline From the American Heart Association/American Stroke Association. Stroke. 2023 Jul;54(7):e314-e370. doi: 10.1161/STR.0000000000000436. Epub 2023 May 22. PMID 37212182
- See also: Ministry of Health webiste — https://www.salute.gov.it/portale/documentazione/p6_2_2_1.jsp?id=959